CLINICAL TRIAL: NCT05280860
Title: Effect of Bilateral Rectus Sheath Block on Postoperative Delirium in Elderly Patients Undergoing Laparoendoscopic Single-site Surgery ：A Prospective, Double-Blind, Randomized, Clinical Trial
Brief Title: Effect of Bilateral RSB on Postoperative Delirium in Elderly Patients Undergoing Laparoendoscopic Single-site Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-k033
Record Dates: First submitted 2021-12-23; First posted 2022-03-15 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2021-12

CONDITIONS: Delirium in Old Age; Hernia, Inguinal; Cholecystolithiasis
MeSH Terms: conditions — Hernia, Inguinal; Cholecystolithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group R: bilateral RSB under ultrasound guidance after general anesthesia (Experimental): Group R was subjected to a bilateral RSB under ultrasound guidance after general anesthesia.
  Interventions: Procedure: ultrasound-guided bilateral rectus sheath block
- Group G: simple general anesthesia (No Intervention): Group G received simple general anesthesia.

INTERVENTIONS:
Procedure: ultrasound-guided bilateral rectus sheath block — Bilateral RSB was guided by ultrasound before surgery after the completion of general anesthesia, First, the probe is placed transversely and perpendicular to reveal the anterior, hypoechoic, and posterior rectus sheath of the hyperechoic rectus abdominis. Moving the probe outward to reveal the sound images of the lateral margin of the rectus abdominis, external oblique, internal oblique, and transverse abdominis muscles. After the scanning, the needle was inserted from any segment of the probe under the guidance of real-time ultrasound; the tip reached between the rectus abdominis muscle and the posterior sheath of the rectus abdominis muscle. After no blood was extracted, 1 ~ 2 ml of normal saline was firstly injected to determine whether the tip position was correct, If the needle tip was correctly positioned, 0.5 % ropivacaine 10 mL of local anesthetic was injected on each side. The same anesthesiologist was performed bilateral RSB under ultrasound guidance.
  Arms: Group R: bilateral RSB under ultrasound guidance after general anesthesia

SUMMARY:
Postoperative delirium is a common complication in clinical surgery. It has been reported that it can increase postoperative morbidity and mortality and lead to decreased functional and cognitive abilities. The aim of this study was to investigate the effect of ultrasound-guided bilateral rectus sheath blocks (RSB) on postoperative delirium in elderly patients undergoing laparoendoscopic single-site surgery (LESS) A double-blind, randomized controlled trial was conducted with 320 patients, aged 65-80 years, ASA I-III, who were scheduled to undergoing LESS in our hospital were selected, the patients divided into Group R and Group G by random number table method, with 160 patients in each group. Group R was subjected to a bilateral RSB under ultrasound guidance after general anesthesia, each side was given 0.5% ropivacaine 10 ml. Group G received simple general anesthesia.

The mini-mental State Examination was used to assess all the patients' primary cognitive status one day before surgery. Perioperative variables were recorded to be compared. The investigators used the visual analog scale to assess patients' pain degree with postoperative, using confusion assessment method to assess whether patients experienced delirium.

DETAILED DESCRIPTION:
1. Study design and setting 320 elderly patients undergoing LESS surgery under general anesthesia (including inguinal hernia and cholecystolithiasis), gender, aged 65-80 years, American Society of Anesthesiologists (ASA) physical status I-II. Exclusion criteria: MMSE of 1 day before surgery < 27, communication and dysfunction (e.g., vision, hearing), cerebrovascular history, local anesthetic allergy, opioid allergy, puncture site infection, abnormal clotting.
2. Subjects Patients were allocated randomly to R group (bilateral rectus abdominis sheath blocks combined with the general anesthesia group) and G group (the simple general anesthesia group) according to computer-generated random number table. All patients and an investigator who was responsible for follow-up during 48 postoperative hours were blinded to the randomization groups. In addition, during preoperative visits, the investigators instructed patients how to use the patient-controlled intravenous analgesia (PCA) device for pain management, as well as how to use the visual analog scale to evaluate pain at rest and while coughing. All the bispectral index (BIS) value in the present study was maintained between 40 and 60 during surgery. All patients voluntarily signed informed consent.
3. General anesthesia Patients were monitored by electrocardiogram, pulse oximetry and non-invasive blood pressure (one measurement every 3 min) while entering operation room. A radial artery catheter was also placed for invasive arterial pressure and blood gas monitoring. The induction of general anaesthesia was performed intravenously with sufentanil 0.5 µg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg. Endotracheal intubation was performed with a double-lumen tube. Sevoflurane was wsed at a minimal alveolar concentration (MAC) of 0.8-1, remifentanil and propofol were used for the maintenance. Fluid management was at the discretion of the attending anaesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 to 80 years male and female
* Scheduled for elective single-incision laparoscopic cholecystectomy
* The patients volunteered to participate in the study and signed the informed consent

Exclusion Criteria:

* Preexisting neuropathy
* Coagulopathy
* Local skin infection
* Hepatic, renal or cardiorespiratory failure
* Local anesthetic allergy
* Pregnancy
* Complications of gallstone with gallbladder perforation
* Diffuse peritonitis
* Acute pyogenic cholangitis

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
The mini-mental State Examination | one day before the operation.
  The mini-mental State Examination is effective as a screening tool for cognitive impairment with older, community dwelling, hospitalized and institutionalized adults. Assessment of an older adult's cognitive function is best achieved when it is done routinely, systematically and thoroughly. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age.
Change from Baseline visual analogue scale | 30 minutes after extubation and 6 hours and 12 hours
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity. Based on the distribution of pain Visual Analogue Scale scores in post-surgical patients (knee replacement, hysterectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain Visual Analogue Scale have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
The effective times of patient-controlled intravenous analgesia | during 0-6 hours, 6-12 hours, and 12-24 hours
  Change from Baseline patient-controlled intravenous analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Principal Investigator — Ethics Committee of Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No